CLINICAL TRIAL: NCT02715544
Title: Promoting Healthy Eating and Active Playtime by Connecting Preschool Children to Nature
Acronym: Play&Grow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Tanja Sobko, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P&G 2015
Record Dates: First submitted 2016-03-08; First posted 2016-03-22 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Sedentary Lifestyle; Overweight; Eating Disorders
Keywords: Intervention; Physical activity; Eating habit; Connectedness to nature
MeSH Terms: conditions — Sedentary Behavior; Overweight; Feeding and Eating Disorders; Motor Activity; Feeding Behavior | interventions — Exercise; Nutrition Policy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): The group will receive healthy lifestyle intervention
  Interventions: Other: Healthy lifestyle
- control group (Active Comparator): Other: physical activity and dietary guidelines
  Interventions: Other: physical activity and dietary guidelines

INTERVENTIONS:
Other: Healthy lifestyle — The families will receive a designed for these purposes intervention
  Arms: Intervention group
Other: physical activity and dietary guidelines — The families will receive a designed for these purposes intervention
  Arms: control group

SUMMARY:
Recent research suggests a majority of Hong Kong's toddlers (aged 2 to 4) are much less active than is recommended and are increasingly engaged in sedentary behaviour, which places them at risk of becoming overweight or obese. The proposed project will test whether connecting families to nature positively influences physical activity (that is, active playtime) and healthy eating routines in children aged 2 to 4. The investigators have recently conducted a pilot study Play & Grow (P&G), a programme based on the most successful international preschool interventions described in the literature. In addition to adopting healthy eating and physical activity intervention elements, the programme was enhanced by including a novel third element: connectedness to nature (CN). To test the effectiveness of this enhanced intervention, the plan is to run a family-based randomised controlled trial (RCT). The intervention will include 240 families with children aged 2 to 4, will take the form of one-hour activity sessions for parents and children held once a week for 10 weeks. The investigators will assess lifestyle-related habits before, immediately after the completion the intervention, at 6 months and one year after the intervention. Created for this purpose, a novel measuring tool for connectedness to nature, Nature Relatedness Scale (NRS), will be validated and tested for reliability prior to the RTC. The results of RCT are intended to be used to understand which components of the intervention were most effective. The objectives of this project will be achieved over a 36-month period, and it is expected to contribute to a close examination of key components of successful healthy lifestyle promotion programme during early childhood. The investigators predict that is that the new element CN will significantly improve the intervention. Finally, the overall aim is that connecting families to nature will result in sustainable lifestyle changes that remain with them for a lifetime.

DETAILED DESCRIPTION:
Proper nutrition and physical activity are essential for a healthy life. Time spent in nature has also been proven beneficial. Systematic reviews have shown that nature-related activities enhance general well-being as reflected in increased physical activity, a healthier diet, reduced stress and better sleep. However, existing programmes promoting healthy lifestyles in children focus almost exclusively on diet and physical activity. None, to the inestigators's awareness, taken into consideration interactions, or connectedness with nature. Connectedness to nature/nature relatedness is a relatively new concept that, to date, has been investigated primarily in adults.The concept suggests, for example, that engaging in activities in a natural environment can induce a feeling of connectedness to nature. Exposing preschool children to nature and to thinking about nature in different ways could stimulate nature relatedness as a measurable construct. When children are placed in a natural setting, they are more likely to be physically active. Natuxral products such as fruits and vegetables are widely acknowledged to improve health. As noted above, parents are children's role models, and the investigators therefore believe that connecting parents with nature will have benefits for their children. Many habits and attitudes are developed early in life, and those related to the natural world are no exception. In fact, children are inherently interested in their environment and in nature in general. The hypothesis is that both indoor and outdoor nature-related activities may induce connectedness and bring about positive changes in both eating and activity habits (short-term outcomes) in preschool children, in turn leading to a healthier lifestyle (long-term outcomes).The aim of P&G is to encourage healthy eating habits and active play in children from an early age, and to bring about healthy behavioural changes in families. The programme also includes a CN element designed to equip parents with environmental knowledge and skills. The generated re- and post-test comparison data indicated the effectiveness of the programme (not presented here). A detailed manual and full resource kit were created, and each session consisted of: (i) a 15-minute theoretical education component (food, activity, CN), and (ii) a 30-minute component on indoor and outdoor nature-related activities, such as playing with nature objects and searching for natural treasures. Some nature activities were food-related (e.g. growing plants, creating miniature indoor gardens, and healthy cooking). The control group received an information folder containing government-recommended physical activity and dietary guidelines for children. To enhance participation, the sessions were scheduled for weekends. The outcome data was collected using a number of scales and questionnaires addressed eating, active play and nature-related habits before and after the program, and focus group discussions were held at the beginning and end of the programme. The programme proved popular amongst participants and the results demonstrated significant positive changes on number of health-related outcomes, such as food habits and caregiver physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* 2-4 year old children
* With English-speaking parents

Exclusion Criteria:

* Children with chronic health conditions
* Families who have recently taken part in a healthy lifestyle promotion programme

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Eating habits | 3 years
  A short validated Eating and Physical Activity Questionnaire (EPAQ)
Physical activity | 3 years
  Physical Activity Questionnaire for Preschool-aged Children (Pre-PAQ®)
Nature relatedness | 3 years
  a short, age-adjusted NRS scale

SECONDARY OUTCOMES:
Parental knowledge of nutrition | 3 years
  Nutrition Knowledge Questionnaire (NKQ)
Parental feeding behaviours | 3 years
  The Preschool Child Feeding Questionnaire (PCFQ)
weight | 3 years
  weight in kilograms
height | 3 years
  height in meters
child neophobia | 3 years
  Pliner's Child Neophobia Scale (PCNS)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja sobko, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Hong Kong Ethics Committee

REFERENCES:
- [Background] Nisbet EK, Zelenski JM. The NR-6: a new brief measure of nature relatedness. Front Psychol. 2013 Nov 1;4:813. doi: 10.3389/fpsyg.2013.00813. eCollection 2013. PMID 24198806
- [Background] Cleland V, Crawford D, Baur LA, Hume C, Timperio A, Salmon J. A prospective examination of children's time spent outdoors, objectively measured physical activity and overweight. Int J Obes (Lond). 2008 Nov;32(11):1685-93. doi: 10.1038/ijo.2008.171. Epub 2008 Oct 14. PMID 18852701
- [Background] Dyment JE, Bell AC. Grounds for movement: green school grounds as sites for promoting physical activity. Health Educ Res. 2008 Dec;23(6):952-62. doi: 10.1093/her/cym059. Epub 2007 Oct 22. PMID 17956885
- [Background] Bell JF, Wilson JS, Liu GC. Neighborhood greenness and 2-year changes in body mass index of children and youth. Am J Prev Med. 2008 Dec;35(6):547-53. doi: 10.1016/j.amepre.2008.07.006. PMID 19000844
- [Background] Veselinovska SS, Osogovska TL: Engagement of Students in Environmental Activities in School. Procedia - Social and Behavioral Sciences 2012, 46:5015-5020.
- [Background] Barratt Hacking E, Barratt R, Scott W: Engaging children: research issues around participation and environmental learning. Environmental Education Research 2007, 13:529-544.
- [Background] Mullis F: Active parenting: an evaluation of two Adlerian parent education programs. Journal of Individual Psychology 1999, 55:225-232.
- [Background] Liefländer AK, Fröhlich G, Bogner FX, Schultz PW: Promoting connectedness with nature through environmental education. Environmental Education Research 2013, 19(3):370-384
- [Background] Cutter-Mackenzie A, Edwards S: Toward a Model for Early Childhood Environmental Education: Foregrounding, Developing, and Connecting Knowledge Through Play-Based Learning. The Journal of Environmental Education 2013, 44(3):195-213.
- [Background] The Biophilia Hypothesis [http://books.google.com/books?hl=nl&lr=&id=qOg3-J0BoGoC&pgis=1]
- [Derived] Sobko T, Brown GTL, Cheng WHG. Does connectedness to nature improve the eating behaviours of pre-schoolers? Emerging evidence from the Play&Grow randomised controlled trial in Hong Kong. Appetite. 2020 Nov 1;154:104781. doi: 10.1016/j.appet.2020.104781. Epub 2020 Jun 30. PMID 32615145
- [Derived] Sobko T, Jia Z, Brown G. Measuring connectedness to nature in preschool children in an urban setting and its relation to psychological functioning. PLoS One. 2018 Nov 29;13(11):e0207057. doi: 10.1371/journal.pone.0207057. eCollection 2018. PMID 30496300
- [Derived] Sobko T, Tse M, Kaplan M. A randomized controlled trial for families with preschool children - promoting healthy eating and active playtime by connecting to nature. BMC Public Health. 2016 Jun 13;16:505. doi: 10.1186/s12889-016-3111-0. PMID 27296723
- See also: Programme promotion video — https://www.youtube.com/watch?v=tAgGCYbPwHs